CLINICAL TRIAL: NCT00177411
Title: "Determining the Maximum Tolerable Dose and Pharmacokinetic Parameters of Intravenous PTHrP(1-36)"
Brief Title: "PTHrP(1-36) IV Dose Escalation Study"
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Protocol design was changed so it no longer fit the description of this study.
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Mara Horwitz, Associate Professor of Medicne, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IRB # 0507001; R01DK051081 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Osteoporosis
Keywords: Endocrine System Diseases; MusculoSkeletal System Diseases; Hormone; Postmenopausal Women
MeSH Terms: conditions — Osteoporosis; Endocrine System Diseases; Musculoskeletal Diseases | interventions — Parathyroid Hormone-Related Protein; parathyroid hormone-related peptide (1-36)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PTHrP group (Experimental): Subjects receiving PTHrP in varying doses.
  Interventions: Drug: Parathyroid Hormone-related Protein

INTERVENTIONS:
Drug: Parathyroid Hormone-related Protein — Parathyroid Hormone-related Protein in doses started at a 4 microgram single bolus intravenous dose. Dose will be increase to a maximum of 400 micrograms or until a dose limiting toxicity occurs at a lower dose.
  Other Names: PTHrP(1-36)

SUMMARY:
This is a single-blinded, one-treatment, combination dose escalation and pharmacokinetic study done in healthy volunteers. The investigators want to determine whether Parathyroid Hormone related Protein (1-36) [PTHrP(1-36)] shares anabolic properties with the only currently approved anabolic agent, parathyroid hormone(1-34) [PTH(1-34)], which stimulates both osteoblastic bone resorption and formation. In a previous study done by the investigators, postmenopausal osteoporotic women on estrogen received 6.56 mcg/kg PTHrP(1-36) subcutaneously for three months daily. They experiences a 4.7% increase in bone mineral density (BMD) of the lumbar spine when compared with those taking placebo. They also displayed an increase in serum osteocalcin, a marker of bone formation, with no change in several markers of bone resorption. It is believed that the rapid absorption and clearance of PTHrP(1-36) likely plays a central role in its anabolic effect In order to further assess absorption, we are combining both pharmacokinetic and dose escalation methods for studying intravenous PTHrP given via a one-time bolus injection. The purpose is to define the maximum safe dose and measure the pharmacokinetic parameters of a single intravenous dose of Parathyroid Hormone-related Protein (1-36)[PTHrP(1-36)]. The results will be useful in determining future treatment options for osteoporosis.

DETAILED DESCRIPTION:
Osteoporosis is a growing health problem. The most commonly used treatment options are anti-resorptive agents, which give a bone density increase of the lumbar spine in the 6-8% range over a 3-5 year period. A 100 % increase in bone mass would be needed to restore bone mass to peak, premenopausal levels. The ideal drug to treat osteoporosis would be a pure skeletal anabolic agent; however, the only currently approved anabolic agent, parathyroid hormone [PTH(1-34)] appears to only increase lumbar spine mass by 12-15% over a 2-3 year period when given alone.

Parathyroid hormone-related protein, [PTHrP(1-36)], is a peptide secreted by almost all normal tissues and cells that shares significant homology with Parathyroid Hormone (PTH); and the investigators believe that it shares anabolic properties with PTH. In a previous study, PTHrP(1-36) administered subcutaneously to postmenopausal women for two weeks increased markers of bone formation (osteocalcin) while decreasing markers of osteoclastic bone resorption. In a subsequent study, postmenopausal osteoporotic women on estrogen received 6.56 mcg/kg PTHrP(1-36) subcutaneously for 3 months daily. They experienced a 4.7% increase in bone mineral density (BMD) of the lumbar spine compared to those taking placebo. The also displayed an increase in serum osteocalcin, a marker of bone formation, with no change in several markers of bone resorption. As a result of both rat and human research studies, the investigators feel the rapid absorption and clearance of PTHrP(1-36) likely plays a central role in its anabolic effect in humans.

In order to further assess the absorption of PTHrP, the investigators are doing this pharmacokinetic study using bolus intravenous PTHrP. It combines both pharmacokinetic and dose escalation methods for studying intravenous PTHrP given via a one-time bolus injection. Subcutaneous PTHrP has been shown to increase bone mass in previous studies done and would be the preferred route for administration of PTHrP in the treatment of osteoporosis. Comparing intravenous with subcutaneous PTHrP will yield much information about the bioavailability of PTHrP in vivo.

This six hour study has been designed to achieve the goals of (1) determining what is the maximum safe dose of PTHrP(1-36) that can be given intravenously as a one time bolus dose; and (2) what is the pharmacokinetic profile of a one-time intravenous bolus dose of PTHrP. A placebo group of 5 subjects will initially serve as a control. The investigators feel it is important to begin with very small amounts of intravenous PTHrP and gradually increase the dose for safety reasons. The initial single bolus intravenous dose to be tested is intentionally low (4 micrograms). Subsequent doses of PTHrP will be gradually increased using a standard dose escalation scale in groups of three subjects until a maximal dose of 400 mcg is reached or a dose limiting toxicity occurs at a dose lower than 400 mcg. The maximum determined safely tolerated dose will then be administered to a total of 10 normal healthy volunteers.

In all subjects at different dosing groups, frequent blood sampling within the first 20 minutes after IV administration of PTHrP will yield pharmacokinetic data about peak PTHrP blood levels and time to peak level T(max). After research subjects receive an intravenous bolus of PTHrP; blood samples will be collected for pharmacokinetic analysis of PTHrP at intervals of 2 minutes for the first 20 minutes, than at 25, 30, 45 and 60 minutes, then hourly for the next five hours. Measurement of calcium, creatinine, phosphorus, PTH, 1,25 Vitamin D and markers of bone metabolism will be obtained at baseline, and at hours one and three. After the baseline urine sample is obtained, urine will be collected at two hour intervals for calcium, creatinine, phosphorus, and markers of bone metabolism.

All subjects will be assigned in a single-blinded manner to receive either placebo or study drug. Initial subjects will be assigned to receive placebo or the starting dose of PTHrP: 4 micrograms. all groups of subjects will receive of PTHrP or placebo via intravenous bolus injection followed by a 3 ml normal saline solution flush over a 30-60 period. If subjects in the initial groups do not experience any adverse effects, doses of intravenous PTHrP will be increased in subsequent groups of three subjects each, and the doses for these groups will be 10, 40, 75, 150, 250 and lastly, 400 micrograms. 400 micrograms is the highest possible dose that will be given in this study. The dose that causes no dose-limiting toxicities will be given to a total of 10 healthy subjects. Data from this dosing group will be used to compare data from the investigator's previous pharmacokinetic and dose escalation studies, including recently completed a double-blind, crossover pharmacokinetic study comparing peak serum levels of PTH(1-34) and PTHrP(1-36) after a single subcutaneous injection. Preliminary results from that study indicated that PTHrP peaks earlier than PTH (6-15 minutes verses 45 minutes), despite the fact that the dose of PTHrP (~420 mcg) was 20 times greater than the dose of PTH (20 mcg).

This study will be performed in healthy young adults, ages 24-35 years. It is anticipated that we will need to screen 100 subjects to achieve a maximum of 52 evaluable subjects, to answer the questions posed by this study.

ELIGIBILITY:
Inclusion Criteria:

Healthy Caucasian subjects of both sexes between the ages of 24-35 years -

Exclusion Criteria:

Pregnancy Subjects with cardiac, hypertension, vascular, renal, pulmonary, endocrine, musculoskeletal, hepatic hematologic or malignant or rheumatologic disease.

Body Mass Index greater than 30 anemia (hematocrit less than 36% in women, less than 40% in men) significant alcohol or drug abuse, baseline hypotension (systolic blood pressure less than 90 mm/HG) baseline hypertension (systolic BP greater than 140 mmHg or diastolic BP greater than 90 mmHg Abnormal screening labs including: ionized and total serum calcium, phosphorus, creatinine, albumin, 25-hydroxyvitamin D, and PTH.

Subjects taking any chronic medication except oral contraceptives Those who have received an investigational drug in the past 90 days Any subject who has previously received either PTH or PTHrP African Americans and other ethnic minorities will be excluded since it is well documented that osteoporosis is far more common in Caucasians than in African-Americans, and there are clear quantitative differences in bone density and sensitivity to parathyroid hormone between African-Americans and Caucasians. -

Ages: 24 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2005-07; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The absence of any dose limiting toxicity criteria | 6 hours

SECONDARY OUTCOMES:
Measurement of vitamin D levels, markers of bone metabolism and fractional excretion of calcium measurements | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mara J. Horwitz, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Horwitz MJ, Tedesco MB, Gundberg C, Garcia-Ocana A, Stewart AF. Short-term, high-dose parathyroid hormone-related protein as a skeletal anabolic agent for the treatment of postmenopausal osteoporosis. J Clin Endocrinol Metab. 2003 Feb;88(2):569-75. doi: 10.1210/jc.2002-021122. PMID 12574182
- [Background] Syed MA, Horwitz MJ, Tedesco MB, Garcia-Ocana A, Wisniewski SR, Stewart AF. Parathyroid hormone-related protein-(1--36) stimulates renal tubular calcium reabsorption in normal human volunteers: implications for the pathogenesis of humoral hypercalcemia of malignancy. J Clin Endocrinol Metab. 2001 Apr;86(4):1525-31. doi: 10.1210/jcem.86.4.7406. PMID 11297578
- [Background] Horwitz MJ, Tedesco MB, Sereika SM, Hollis BW, Garcia-Ocana A, Stewart AF. Direct comparison of sustained infusion of human parathyroid hormone-related protein-(1-36) [hPTHrP-(1-36)] versus hPTH-(1-34) on serum calcium, plasma 1,25-dihydroxyvitamin D concentrations, and fractional calcium excretion in healthy human volunteers. J Clin Endocrinol Metab. 2003 Apr;88(4):1603-9. doi: 10.1210/jc.2002-020773. PMID 12679445
- [Background] Everhart-Caye M, Inzucchi SE, Guinness-Henry J, Mitnick MA, Stewart AF. Parathyroid hormone (PTH)-related protein(1-36) is equipotent to PTH(1-34) in humans. J Clin Endocrinol Metab. 1996 Jan;81(1):199-208. doi: 10.1210/jcem.81.1.8550752.
- [Background] Henry JG, Mitnick M, Dann PR, Stewart AF. Parathyroid hormone-related protein-(1-36) is biologically active when administered subcutaneously to humans. J Clin Endocrinol Metab. 1997 Mar;82(3):900-6. doi: 10.1210/jcem.82.3.3811. PMID 9062504
- [Background] Plotkin H, Gundberg C, Mitnick M, Stewart AF. Dissociation of bone formation from resorption during 2-week treatment with human parathyroid hormone-related peptide-(1-36) in humans: potential as an anabolic therapy for osteoporosis. J Clin Endocrinol Metab. 1998 Aug;83(8):2786-91. doi: 10.1210/jcem.83.8.5047. PMID 9709948
- [Background] Stewart AF, Cain RL, Burr DB, Jacob D, Turner CH, Hock JM. Six-month daily administration of parathyroid hormone and parathyroid hormone-related protein peptides to adult ovariectomized rats markedly enhances bone mass and biomechanical properties: a comparison of human parathyroid hormone 1-34, parathyroid hormone-related protein 1-36, and SDZ-parathyroid hormone 893. J Bone Miner Res. 2000 Aug;15(8):1517-25. doi: 10.1359/jbmr.2000.15.8.1517. PMID 10934650
- [Background] Bisello A, Horwitz MJ, Stewart AF. Parathyroid hormone-related protein: an essential physiological regulator of adult bone mass. Endocrinology. 2004 Aug;145(8):3551-3. doi: 10.1210/en.2004-0509. No abstract available. PMID 15265822
- [Background] Horwitz MJ, Tedesco MB, Sereika SM, Syed MA, Garcia-Ocana A, Bisello A, Hollis BW, Rosen CJ, Wysolmerski JJ, Dann P, Gundberg C, Stewart AF. Continuous PTH and PTHrP infusion causes suppression of bone formation and discordant effects on 1,25(OH)2 vitamin D. J Bone Miner Res. 2005 Oct;20(10):1792-803. doi: 10.1359/JBMR.050602. Epub 2005 Jun 6. PMID 16160737
- [Background] Horwitz MJ, Tedesco MB, Sereika SM, Garcia-Ocana A, Bisello A, Hollis BW, Gundberg C, Stewart AF. Safety and tolerability of subcutaneous PTHrP(1-36) in healthy human volunteers: a dose escalation study. Osteoporos Int. 2006 Feb;17(2):225-30. doi: 10.1007/s00198-005-1976-3. Epub 2005 Sep 7. PMID 16151606